CLINICAL TRIAL: NCT07068204
Title: Caries-preventing Effect of 2% Calcium Hypophosphite Toothpaste Compared to a Sodium Fluoride Toothpaste (1450ppm F) in Adults
Brief Title: Comparative Study of Caries-Preventive Effects: 2% Calcium Hypophosphite Toothpaste vs. Sodium Fluoride Toothpaste (1450ppm F)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Joachim Enax (Industry)
Collaborators: Department of Integrated Dentistry Medical University of Białystok (Unknown); Poznan University of Medical Sciences, Department of Integrated Dentistry (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Joachim Enax, Senior Scientist Oral Care, Dr. Kurt Wolff GmbH & Co. KG
Organization: Dr. Kurt Wolff GmbH & Co. KG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CA2-04/2024
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Caries, Dental; Calcium Hypophosphite; Fluoridation
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2% Calcium Hypophosphite Toothpaste (Experimental)
  Interventions: Device: 2% Calcium Hypophosphite Toothpaste
- Sodium Fluoride Toothpaste (1450 ppm F) (Placebo Comparator)
  Interventions: Device: Sodium Fluoride Toothpaste (1450 ppm F)

INTERVENTIONS:
Device: 2% Calcium Hypophosphite Toothpaste — Oral hygiene instruction and regular application of the 2% Calcium Hypophosphite Toothpaste at home (twice daily over a period of 546 days, i.e., 18 months).
  Arms: 2% Calcium Hypophosphite Toothpaste
Device: Sodium Fluoride Toothpaste (1450 ppm F) — Oral hygiene instruction and regular application of the Sodium Fluoride Toothpaste at home (twice daily over a period of 546 days, i.e., 18 months).
  Arms: Sodium Fluoride Toothpaste (1450 ppm F)

SUMMARY:
The aim of the study is to compare the caries-preventive effect of the test and control toothpaste in order to proof the non-inferiority of the test toothpaste compared to the control.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 10 healthy molars and premolars (DMFS of these teeth = 0)
* Willingness to use an electric (powered) toothbrush
* Willingness to use interdental floss
* Willingness to have bitewing radiographs taken
* Willingness to undergo an oral examination by an intraoral camera (DIAGNOcam)

Exclusion Criteria:

* Untreated caries [clinical investigation and analysis with an intraoral camera (DIAGNOcam)] (→ unsuitable subjects with one or two untreated caries in need of a restoration can become eligible after restorative therapy. If there are three or more untreated caries patients will be excluded)
* Xerostomia (medication, radiation, disease induced)
* Chemo/radiation therapy
* Physical or mental disability which prevents proper oral health care
* Orthodontic treatment
* Severe periodontitis at the Baseline Visit (pocket depth on at least one tooth ≥ 5.5 mm)
* Known hypersensitivity to one of the ingredients of the toothpastes to be tested
* Regular medication intake interfering with salivary function or flow
* Current pregnancy, the wish to become pregnant, the suspicion of being pregnant, or breastfeeding or in the course of the study
* 3 or more carious lesions/restorations in last 36 months until Baseline Visit
* Teeth missing due to caries in last 36 months until Baseline Visit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of the 2% Calcium Hypophosphite Toothpaste compared to Sodium Fluoride Toothpaste (1450 ppm F) regarding the Decay-Missing-Filled index | Day 1, Day 182±28, Day 365±28 vs. Day 546±28
  Comparison between the 2% Calcium Hypophosphite Toothpaste and Sodium Fluoride Toothpaste (1450 ppm F): Proportion of subjects showing no increase in overall Decay-Missing-Filled index during the observation period of 546 days (assessed by the investigator).

SECONDARY OUTCOMES:
Evaluate the efficacy of the 2% Calcium Hypophosphite Toothpaste compared to Sodium Fluoride Toothpaste (1450 ppm F) in the prevention of interproximal caries lesions | Day 1 vs. Day 546±28
  Comparison between 2% Calcium Hypophosphite Toothpaste and Sodium Fluoride Toothpaste (1450 ppm F): Proportion of subjects with no change in mineral density, as analyzed by DIAGNOcam Full Vision HD using near-infrared laser transillumination, over an observation period of 546 days (assessed by the investigator).
Evaluate the efficacy of 2% Calcium Hypophosphite Toothpaste compared to Sodium Fluoride Toothpaste (1450 ppm F) in the prevention of dental plaque deposition using the Plaque Control Record (PCR) index | Day 1, Day 182±28, Day 365±28 vs. Day 546±28
  At the study visits, a suitable disclosing solution such as Bismarck Brown, Diaplac or similar is painted on tooth surfaces. After the subject has rinsed, the investigator (using an explorer or a tip of a probe) examines each stained surface for soft accumulations at the dentogingival junction. After all teeth have been examined and scored, the index is calculated by dividing the number of plaque containing surfaces by the total number of available surfaces.
  Plaque Control Record Index Calculation = The number of plaque containing surfaces / The total number of available surfaces

CONTACTS AND LOCATIONS:
Overall Officials: Elzbieta Paszynska, Prof., DDS, Msc, PhD, Principal Investigator — Poznan University of Medical Sciences; Malgorzata Pawinska, Assoc. Prof., DDS, PhD, Principal Investigator — Department of Integrated Dentistry Medical University of Białystok

IPD SHARING:
Plan to Share IPD: No